CLINICAL TRIAL: NCT01591460
Title: An International, Multicenter, Open-Label Study Evaluating Sustained Virological Response and Safety With Boceprevir in Triple Combination Therapy With Peginterferon Alfa-2a (40KD) and Ribavirin in Treatment-Naïve Patients With Genotype 1 Chronic Hepatitis C
Brief Title: A Triple Combination Therapy Study of Boceprevir, Pegasys and Copegus in Previously Untreated Patients With Genotype 1 Chronic Hepatitis C
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MV28073; 2011-004810-41 (EudraCT Number)
Record Dates: First submitted 2012-05-02; First posted 2012-05-04 (Estimated); Results first posted 2015-08-07 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Hepatitis C, Chronic
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — N-(3-amino-1-(cyclobutylmethyl)-2,3-dioxopropyl)-3-(2-((((1,1-dimethylethyl)amino)carbonyl)amino)-3,3-dimethyl-1-oxobutyl)-6,6-dimethyl-3-azabicyclo(3.1.0)hexan-2-carboxamide; peginterferon alfa-2a; Ribavirin

ARMS (2):
- Dual Combination Therapy (Experimental)
  Interventions: Drug: peginterferon alfa-2a [Pegasys]; Drug: ribavirin (Copegus]
- Triple Combination Therapy (Experimental)
  Interventions: Drug: boceprevir; Drug: peginterferon alfa-2a [Pegasys]; Drug: ribavirin (Copegus]

INTERVENTIONS:
Drug: boceprevir — 800 mg three times daily for 24, 32 or 44 weeks
  Arms: Triple Combination Therapy
Drug: peginterferon alfa-2a [Pegasys] — 180 mcg subcutaneously once a week for 24, 32 or 44 weeks
  Arms: Triple Combination Therapy
Drug: peginterferon alfa-2a [Pegasys] — 180 mcg subcutaneously once a week for 4 weeks
  Arms: Dual Combination Therapy
Drug: ribavirin (Copegus] — 1000 mg or 1200 mg orally once a day for 24, 32 or 44 weeks
  Arms: Triple Combination Therapy
Drug: ribavirin (Copegus] — 1000 mg or 1200 mg orally once a day for 4 weeks
  Arms: Dual Combination Therapy

SUMMARY:
This open-label, multicenter, treatment response guided study will evaluate the sustained virological response and safety of the triple combination therapy boceprevir, Pegasys (peginterferon alfa-2a) and Copegus (Ribavirin) in previously untreated patients with genotype 1 chronic hepatitis C. In the lead-in phase, patients will receive a dual combination therapy of Pegasys and Copegus for 4 weeks. In the following triple combination therapy phase, 800 mg boceprevir, 180 mcg Pegasys and 1000-1200 mg Copegus will be administered for 24, 32 or 44 weeks; the duration depending on the patient's treatment response. The anticipated time on study treatment is up to 48 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients >/=18 years of age
* Chronic liver disease consistent with chronic hepatitis C, genotype 1 infection
* Serum HCV RNA quantifiable at screening
* Patients who have not been previously treated with pegylated interferon (IFN), standard IFN, RBV or any direct acting anti-viral agent
* Compensated liver disease (Child-Pugh Grade A clinical classification for patients with cirrhosis: total score </=6)
* Negative urine or blood pregnancy test (for women of childbearing potential)

Exclusion Criteria:

* Women with ongoing pregnancy or breast feeding
* Male partners of women who are pregnant
* Therapy with any systemic anti-viral, anti-neoplastic or immunomodulatory treatment </=6 months prior to the first dose of study drug
* Any investigational drug </=6 weeks prior to the first dose of study drug
* History or other evidence of decompensated liver disease
* History or other evidence of a medical condition associated with chronic liver disease other than chronic hepatitis C
* Signs or symptoms of hepatocellular carcinoma
* Co-infection with HCV genotypes other than genotype 1
* Co-infection with hepatitis A, hepatitis B, and/or human immunodeficiency virus (HIV)
* Any patient with an increased risk for anemia
* History of severe psychiatric disease
* History of immunologically mediated, chronic pulmonary, or severe cardiac disease
* Current diseases that are not adequately controlled

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Actual)
Dates: Start 2012-08; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (26):
- Austria (4):
  - Graz
  - Innsbruck
  - Linz
  - Vienna
- Germany (5):
  - Dortmund
  - Frankfurt am Main
  - Hamburg
  - Hanover
  - Oberhausen
- Hungary (4):
  - Budapest
  - Debrecen
  - Kaposvár
  - Pécs
- Poland (6):
  - Bialystok
  - Bydgoszcz
  - Chorzów
  - Lodz
  - Lublin
  - Wroclaw
- Romania (3):
  - Bucharest
  - Constanța
  - Timișoara
- Spain (4):
  - Granada, Granada
  - Vigo, Pontevedra
  - Barakaldo, Vizcaya
  - Zaragoza, Zaragoza

REFERENCES:
- [Derived] Ferenci P, Caruntu FA, Lengyel G, Messinger D, Bakalos G, Flisiak R. Boceprevir Plus Peginterferon Alfa-2a/Ribavirin in Treatment-Naive Hepatitis C Virus Genotype 1 Patients: International Phase IIIb/IV TriCo Trial. Infect Dis Ther. 2016 Jun;5(2):113-24. doi: 10.1007/s40121-016-0110-5. Epub 2016 May 26. PMID 27228998

RESULTS

PARTICIPANT FLOW:
Groups:
- Total Population: Treatment-naive participants with chronic hepatitis C (CHC) received treatment with peginterferon alfa-2a (PEG-IFN) 180 micrograms (mcg) subcutaneous (SC) once weekly, weight-based ribavirin (RBV) 1000 to 1200 milligrams (mg) orally (PO) daily in 2 divided doses, and boceprevir 800 mg PO every 7 to 9 hours. Participants received dual therapy with PEG-IFN and RBV from Week 0 to 4, and triple therapy was initiated at Week 4. Those with undetectable hepatitis C virus (HCV) ribonucleic acid (RNA) at Weeks 8 and 24 stopped treatment at Week 28. Those with detectable HCV RNA at Week 8 but undetectable HCV RNA at Week 24 continued triple therapy until Week 36 and received dual therapy from Week 36 to 48. Those with a less than (<) 1-log decrease in HCV RNA at Week 4 continued triple therapy until Week 48, with optional dual therapy from Week 32 to 48 if triple therapy was not tolerated. Participants with compensated cirrhosis, regardless of response, received triple therapy until Week 48.
Period: Overall Study
Arm/Group | Total Population
Started | 165 (Those with elevated (Week 12) or detectable (Week 24) virus discontinued due to the Futility Rule.)
Completed | 139 (The number who completed PEG-IFN, as scheduled according to response-guided treatment, is presented.)
Not Completed | 26
Not completed — Adverse Event or Intercurrent Illness | 5
Not completed — Futility Rule (Week 12) | 7
Not completed — Futility Rule (Week 24) | 3
Not completed — Rebound or Breakthrough | 3
Not completed — Treatment Discontinued by Error | 1
Not completed — Lost to Follow-up | 1
Not completed — Noncompliance | 1
Not completed — Participant Refusal | 3
Not completed — Withdrawal by Subject | 1
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Population: All-Treated Population: All enrolled participants who received at least one dose of study medication.
Groups:
- Total Population: Treatment-naive participants with CHC received treatment with PEG-IFN 180 mcg SC once weekly, weight-based RBV 1000 to 1200 mg PO daily in 2 divided doses, and boceprevir 800 mg PO every 7 to 9 hours. Participants received dual therapy with PEG-IFN and RBV from Week 0 to 4, and triple therapy was initiated at Week 4. Those with undetectable HCV RNA at Weeks 8 and 24 stopped treatment at Week 28. Those with detectable HCV RNA at Week 8 but undetectable HCV RNA at Week 24 continued triple therapy until Week 36 and received dual therapy from Week 36 to 48. Those with a <1-log decrease in HCV RNA at Week 4 continued triple therapy until Week 48, with optional dual therapy from Week 32 to 48 if triple therapy was not tolerated. Participants with compensated cirrhosis, regardless of response, received triple therapy until Week 48.
Arm/Group | Total Population
Number analyzed (Participants) | 165
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.8 (12.53)
Gender [Count of Participants; unit: Participants]
  Female | 83
  Male | 82

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Sustained Virological Response (SVR) at 12 Weeks After End of Treatment (EOT)
Description: SVR at 12 weeks after EOT was defined as an undetectable HCV RNA viral load obtained 12 weeks following completion of treatment. HCV RNA viral load was measured using the Roche COBAS TaqMan 2.0 HCV Test, with a lower limit of detection (LOD) of 10 to 15 international units per milliliter (IU/mL). The percentage of participants with SVR was calculated as [number of participants with undetectable HCV RNA at 12 weeks after EOT divided by the number of participants analyzed] multiplied by 100.
Time Frame: At 12 weeks after EOT (up to 60 weeks)
Population: All-Treated Population. Arms were not mutually exclusive.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Cirrhotics: Treatment-naive participants with CHC received treatment with PEG-IFN 180 mcg SC once weekly, weight-based RBV 1000 to 1200 mg PO daily in 2 divided doses, and boceprevir 800 mg PO every 7 to 9 hours. Participants received dual therapy with PEG-IFN and RBV from Week 0 to 4, and triple therapy was initiated at Week 4. Response-guided treatment was determined by assessments of virologic response at Weeks 4, 8, and 24. Participants with compensated cirrhosis (Cirrhotics), regardless of response, received triple therapy until Week 48.
- Poor Responders: Treatment-naive participants with CHC received treatment with PEG-IFN 180 mcg SC once weekly, weight-based RBV 1000 to 1200 mg PO daily in 2 divided doses, and boceprevir 800 mg PO every 7 to 9 hours. Participants received dual therapy with PEG-IFN and RBV from Week 0 to 4, and triple therapy was initiated at Week 4. Response-guided treatment was determined by assessments of virologic response at Weeks 4, 8, and 24. Those without cirrhosis and with a <1-log decrease in HCV RNA at Week 4 (Poor Responders) continued triple therapy until Week 48, with optional dual therapy from Week 32 to 48 if triple therapy was not tolerated.
- Late Responders: Treatment-naive participants with CHC received treatment with PEG-IFN 180 mcg SC once weekly, weight-based RBV 1000 to 1200 mg PO daily in 2 divided doses, and boceprevir 800 mg PO every 7 to 9 hours. Participants received dual therapy with PEG-IFN and RBV from Week 0 to 4, and triple therapy was initiated at Week 4. Response-guided treatment was determined by assessments of virologic response at Weeks 4, 8, and 24. Those without cirrhosis and with detectable HCV RNA at Week 8 but undetectable HCV RNA at Week 24 (Late Responders) continued triple therapy until Week 36 and received dual therapy from Week 36 to 48.
- Early Responders: Treatment-naive participants with CHC received treatment with PEG-IFN 180 mcg SC once weekly, weight-based RBV 1000 to 1200 mg PO daily in 2 divided doses, and boceprevir 800 mg PO every 7 to 9 hours. Participants received dual therapy with PEG-IFN and RBV from Week 0 to 4, and triple therapy was initiated at Week 4. Response-guided treatment was determined by assessments of virologic response at Weeks 4, 8, and 24. Those without cirrhosis and with undetectable HCV RNA at Weeks 8 and 24 (Early Responders) stopped treatment at Week 28.
- Others: Treatment-naive participants with CHC received treatment with PEG-IFN 180 mcg SC once weekly, weight-based RBV 1000 to 1200 mg PO daily in 2 divided doses, and boceprevir 800 mg PO every 7 to 9 hours. Participants received dual therapy with PEG-IFN and RBV from Week 0 to 4, and triple therapy was initiated at Week 4. Response-guided treatment was determined by assessments of virologic response at Weeks 4, 8, and 24. Those not meeting criteria for the other treatment groups (Cirrhotics, Poor Responders, Late Responders, or Early Responders) were classified separately (as Others) and were not treated per response-guided therapy.
Arm/Group | Total Population | Cirrhotics | Poor Responders | Late Responders | Early Responders | Others
Number analyzed (Participants) | 165 | 20 | 24 | 24 | 78 | 19
percentage of participants | 81 [74 to 86] | 70 [46 to 88] | 75 [53 to 90] | 88 [68 to 97] | 95 [87 to 99] | 32 [13 to 57]

2. Secondary Outcome: Percentage of Participants With SVR at 24 Weeks After EOT
Description: SVR at 24 weeks after EOT was defined as an undetectable HCV RNA viral load obtained 24 weeks following completion of treatment. HCV RNA viral load was measured using the Roche COBAS TaqMan 2.0 HCV Test, with a lower LOD of 10 to 15 IU/mL. The percentage of participants with SVR was calculated as [number of participants with undetectable HCV RNA at 24 weeks after EOT divided by the number of participants analyzed] multiplied by 100.
Time Frame: At 24 weeks after EOT (up to 72 weeks)
Population: All-Treated Population. Arms were not mutually exclusive.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Total Population | Cirrhotics | Poor Responders | Late Responders | Early Responders | Others
Number analyzed (Participants) | 165 | 20 | 24 | 24 | 78 | 19
percentage of participants | 80 [73 to 86] | 70 [46 to 88] | 71 [49 to 87] | 88 [68 to 97] | 95 [87 to 99] | 32 [13 to 57]

3. Secondary Outcome: HCV RNA Levels
Description: HCV RNA levels were obtained routinely during and after treatment. Mean HCV RNA levels were calculated by averaging the HCV RNA levels among all participants analyzed at each collection timepoint and expressed in log10 IU/mL.
Time Frame: At Baseline; Weeks 2, 4, 6, 8, 12, 16, 24, 28, and 36; EOT; and 12 and 24 weeks after EOT (up to 72 weeks)
Population: All-Treated Population; number (n) = number of participants who provided evaluable data at the respective visit. Arms were not mutually exclusive.
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | Total Population | Cirrhotics | Poor Responders | Late Responders | Early Responders | Others
Number analyzed (Participants) | 165 | 20 | 24 | 24 | 78 | 19
log10 IU/mL
  Baseline (n=165,20,24,24,78,19) | 6.29 (0.722) | 6.34 (0.710) | 6.40 (0.592) | 6.46 (0.530) | 6.18 (0.796) | 6.34 (0.762)
  Week 2 (n=159,18,24,23,76,18) | 4.86 (1.418) | 5.06 (1.288) | 6.07 (0.610) | 5.38 (0.767) | 4.27 (1.441) | 4.90 (1.597)
  Week 4 (n=158,20,24,22,75,17) | 4.06 (1.525) | 4.30 (1.533) | 5.78 (0.550) | 4.60 (0.874) | 3.25 (1.289) | 4.24 (1.689)
  Week 6 (n=151,18,24,21,73,15) | 1.75 (0.882) | 2.01 (1.002) | 2.70 (0.972) | 1.91 (0.570) | 1.25 (0.154) | 2.18 (1.337)
  Week 8 (n=160,20,24,24,77,15) | 1.47 (0.638) | 1.69 (0.650) | 1.95 (0.874) | 1.52 (0.329) | 1.18 (0.000) | 1.84 (1.236)
  Week 12 (n=160,20,24,24,77,15) | 1.35 (0.682) | 1.41 (0.393) | 1.69 (1.316) | 1.25 (0.107) | 1.18 (0.000) | 1.74 (1.292)
  Week 16 (n=156,19,22,24,78,13) | 1.25 (0.405) | 1.34 (0.459) | 1.46 (0.906) | 1.19 (0.045) | 1.18 (0.000) | 1.32 (0.458)
  Week 24 (n=152,17,23,24,78,10) | 1.41 (1.042) | 1.80 (1.753) | 1.83 (1.696) | 1.18 (0.000) | 1.18 (0.000) | 2.21 (1.916)
  Week 28 (n=143,15,19,23,76,10) | 1.23 (0.480) | 1.18 (0.000) | 1.45 (1.173) | 1.18 (0.000) | 1.18 (0.025) | 1.48 (0.822)
  Week 36 (n=71,16,21,24,3,7) | 1.69 (1.563) | 1.54 (1.412) | 2.00 (2.069) | 1.33 (0.745) | 2.60 (2.466) | 1.91 (1.930)
  EOT (n=162,20,24,23,78,17) | 1.52 (1.120) | 1.58 (1.167) | 1.87 (1.563) | 1.38 (0.996) | 1.18 (0.025) | 2.73 (1.943)
  12 weeks after EOT (n=152,19,24,23,74,12) | 1.92 (1.792) | 2.53 (2.340) | 2.48 (2.345) | 1.48 (1.087) | 1.40 (0.946) | 3.83 (2.789)
  24 weeks after EOT (n=159,20,23,24,78,14) | 2.00 (1.874) | 2.66 (2.351) | 2.39 (2.327) | 1.77 (1.605) | 1.42 (1.053) | 4.05 (2.592)

4. Secondary Outcome: Percentage of Participants With Virological Response
Description: HCV RNA levels were obtained routinely during and after treatment. The percentage of participants with undetectable HCV RNA viral load (ie, virological response) was calculated as [number of participants with undetectable HCV RNA at each timepoint divided by the number of participants analyzed] multiplied by 100.
Time Frame: At Weeks 2, 4, 6, 8, 12, 16, 24, 28, and 36; and EOT (up to 48 weeks)
Population: All-Treated Population. Arms were not mutually exclusive.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Total Population | Cirrhotics | Poor Responders | Late Responders | Early Responders | Others
Number analyzed (Participants) | 165 | 20 | 24 | 24 | 78 | 19
percentage of participants
  Week 2 | 4 [1 to 8] | 0 [0 to 17] | 0 [0 to 14] | 0 [0 to 14] | 6 [2 to 14] | 5 [0 to 26]
  Week 4 | 7 [4 to 12] | 0 [0 to 17] | 0 [0 to 14] | 0 [0 to 14] | 14 [7 to 24] | 5 [0 to 26]
  Week 6 | 41 [34 to 49] | 35 [15 to 59] | 0 [0 to 14] | 4 [0 to 21] | 71 [59 to 80] | 26 [9 to 51]
  Week 8 | 61 [53 to 68] | 45 [23 to 68] | 13 [3 to 32] | 0 [0 to 14] | 100 [95 to 100] | 53 [29 to 76]
  Week 12 | 82 [75 to 87] | 65 [41 to 85] | 75 [53 to 90] | 67 [45 to 84] | 100 [95 to 100] | 53 [29 to 76]
  Week 16 | 87 [81 to 91] | 70 [46 to 88] | 71 [49 to 87] | 96 [79 to 100] | 100 [95 to 100] | 58 [33 to 80]
  Week 24 | 88 [82 to 92] | 80 [56 to 94] | 79 [58 to 93] | 100 [86 to 100] | 100 [95 to 100] | 42 [20 to 67]
  Week 28 | 87 [81 to 91] | 80 [56 to 94] | 79 [58 to 93] | 96 [79 to 100] | 99 [93 to 100] | 42 [20 to 67]
  Week 36 | 83 [76 to 88] | 75 [51 to 91] | 75 [53 to 90] | 96 [79 to 100] | 95 [87 to 99] | 37 [16 to 62]
  EOT | 87 [81 to 92] | 80 [56 to 94] | 79 [58 to 93] | 96 [79 to 100] | 99 [93 to 100] | 47 [24 to 71]

5. Secondary Outcome: Percentage of Participants With at Least a 1-Log, 2-Log, or 3-Log Reduction in HCV RNA
Description: HCV RNA levels were obtained routinely during and after treatment. Reductions in HCV RNA viral load by 1-log, 2-log, or 3-log increments were determined relative to Baseline HCV RNA. Each increment represents a reduction greater than or equal to (≥) the specified log value, including results for which HCV RNA was below the limit of quantification (25 IU/mL). The percentage of participants with each log reduction in HCV RNA was calculated as [number of participants with log reduction divided by the number of participants analyzed] multiplied by 100.
Time Frame: At Weeks 2, 4, 6, 8, 12, 16, 24, and 28
Population: All-Treated Population. Arms were not mutually exclusive.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Total Population | Cirrhotics | Poor Responders | Late Responders | Early Responders | Others
Number analyzed (Participants) | 165 | 20 | 24 | 24 | 78 | 19
percentage of participants
  3-log, Week 2 | 12 [7 to 17] | 5 [0 to 25] | 0 [0 to 14] | 0 [0 to 14] | 19 [11 to 30] | 16 [3 to 40]
  3-log, Week 4 | 29 [22 to 37] | 20 [6 to 44] | 0 [0 to 14] | 8 [1 to 27] | 47 [36 to 59] | 26 [9 to 51]
  3-log, Week 6 | 88 [82 to 92] | 85 [62 to 97] | 75 [53 to 90] | 92 [73 to 99] | 97 [91 to 100] | 63 [38 to 84]
  3-log, Week 8 | 93 [88 to 97] | 95 [75 to 100] | 83 [63 to 95] | 100 [86 to 100] | 100 [95 to 100] | 68 [43 to 87]
  3-log, Week 12 | 95 [91 to 98] | 100 [83 to 100] | 88 [68 to 97] | 100 [86 to 100] | 100 [95 to 100] | 74 [49 to 91]
  3-log, Week 16 | 94 [89 to 97] | 95 [75 to 100] | 88 [68 to 97] | 100 [86 to 100] | 100 [95 to 100] | 68 [43 to 87]
  3-log, Week 24 | 90 [84 to 94] | 80 [56 to 94] | 83 [63 to 95] | 100 [86 to 100] | 100 [95 to 100] | 53 [29 to 76]
  3-log, Week 28 | 88 [83 to 93] | 80 [56 to 94] | 79 [58 to 93] | 96 [79 to 100] | 100 [95 to 100] | 53 [29 to 76]
  2-log, Week 2 | 27 [20 to 34] | 20 [6 to 44] | 0 [0 to 14] | 8 [1 to 27] | 42 [31 to 54] | 26 [9 to 51]
  2-log, Week 4 | 51 [43 to 59] | 50 [27 to 73] | 0 [0 to 14] | 33 [16 to 55] | 76 [65 to 85] | 37 [16 to 62]
  2-log, Week 6 | 95 [90 to 97] | 95 [75 to 100] | 96 [79 to 100] | 96 [79 to 100] | 99 [93 to 100] | 74 [49 to 91]
  2-log, Week 8 | 97 [93 to 99] | 100 [83 to 100] | 100 [86 to 100] | 100 [86 to 100] | 100 [95 to 100] | 74 [49 to 91]
  2-log, Week 12 | 95 [91 to 98] | 100 [83 to 100] | 88 [68 to 97] | 100 [86 to 100] | 100 [95 to 100] | 74 [49 to 91]
  2-log, Week 16 | 94 [89 to 97] | 95 [75 to 100] | 88 [68 to 97] | 100 [86 to 100] | 100 [95 to 100] | 68 [43 to 87]
  2-log, Week 24 | 90 [84 to 94] | 80 [56 to 94] | 83 [63 to 95] | 100 [86 to 100] | 100 [95 to 100] | 53 [29 to 76]
  2-log, Week 28 | 88 [83 to 93] | 80 [56 to 94] | 79 [58 to 93] | 96 [79 to 100] | 100 [95 to 100] | 53 [29 to 76]
  1-log, Week 2 | 55 [47 to 62] | 60 [36 to 81] | 0 [0 to 14] | 54 [33 to 74] | 73 [62 to 82] | 42 [20 to 67]
  1-log, Week 4 | 81 [74 to 86] | 75 [51 to 91] | 0 [0 to 14] | 100 [86 to 100] | 100 [95 to 100] | 84 [60 to 97]
  1-log, Week 6 | 98 [94 to 99] | 95 [75 to 100] | 100 [86 to 100] | 100 [86 to 100] | 100 [95 to 100] | 84 [60 to 97]
  1-log, Week 8 | 98 [95 to 100] | 100 [83 to 100] | 100 [86 to 100] | 100 [86 to 100] | 100 [95 to 100] | 84 [60 to 97]
  1-log, Week 12 | 96 [92 to 99] | 100 [83 to 100] | 96 [79 to 100] | 100 [86 to 100] | 100 [95 to 100] | 74 [49 to 91]
  1-log, Week 16 | 94 [89 to 97] | 95 [75 to 100] | 88 [68 to 97] | 100 [86 to 100] | 100 [95 to 100] | 68 [43 to 87]
  1-log, Week 24 | 91 [85 to 95] | 80 [56 to 94] | 88 [68 to 97] | 100 [86 to 100] | 100 [95 to 100] | 58 [33 to 80]
  1-log, Week 28 | 88 [83 to 93] | 80 [56 to 94] | 79 [58 to 93] | 96 [79 to 100] | 100 [95 to 100] | 53 [29 to 76]

6. Secondary Outcome: Percentage of Participants With Virological Relapse Following EOT Response
Description: Virological relapse was defined as a detectable post-treatment HCV RNA viral load following a previously undetectable EOT level (ie, virological response). The percentage of participants with virological relapse was calculated as [number of participants meeting the above criteria divided by the number of participants analyzed] multiplied by 100.
Time Frame: Up to 72 weeks (at 12 and 24 weeks after EOT)
Population: All-Treated Population; only participants with a previous EOT virological response were included in the analysis. Arms were not mutually exclusive.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Total Population | Cirrhotics | Poor Responders | Late Responders | Early Responders | Others
Number analyzed (Participants) | 143 | 16 | 19 | 23 | 77 | 8
percentage of participants | 7 [3 to 12] | 13 [2 to 38] | 5 [0 to 26] | 9 [1 to 28] | 4 [1 to 11] | 25 [3 to 65]

7. Secondary Outcome: Percentage of Participants With Virological Breakthrough Following On-Treatment Response
Description: Virological breakthrough was defined as an HCV RNA viral load greater than (>) 1000 IU/mL following a previously undetectable level at any time during treatment (ie, virological response). Participants who ultimately achieved an EOT response were not considered for virological breakthrough. The percentage of participants with virological breakthrough was calculated as [number of participants meeting the above criteria divided by the number of participants analyzed] multiplied by 100.
Time Frame: Up to 48 weeks (at Baseline; Weeks 2, 4, 6, 8, 12, 16, 24, 28, and 36; and EOT)
Population: All-Treated Population; only participants with a previous on-treatment virological response were included in the analysis. Arms were not mutually exclusive.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Total Population | Cirrhotics | Poor Responders | Late Responders | Early Responders | Others
Number analyzed (Participants) | 151 | 17 | 19 | 24 | 78 | 13
percentage of participants | 3 [1 to 7] | 0 [0 to 20] | 0 [0 to 18] | 4 [0 to 21] | 0 [0 to 5] | 23 [5 to 54]

8. Secondary Outcome: Percentage of Participants With Virological Rebound Following On-Treatment Decline in HCV RNA
Description: Virological rebound was defined as an HCV RNA viral load >1000 IU/mL and a ≥1-log increase from nadir following a decline in HCV RNA from Baseline at any time during treatment (ie, on-treatment decline). Participants who ultimately achieved an EOT response were not considered for virological rebound. The percentage of participants with virological rebound was calculated as [number of participants meeting the above criteria divided by the number of participants analyzed] multiplied by 100.
Time Frame: Up to 48 weeks (at Baseline; Weeks 2, 4, 6, 8, 12, 16, 24, 28, and 36; and EOT)
Population: All-Treated Population; only participants with a previous on-treatment decline in HCV RNA were included in the analysis. Arms were not mutually exclusive.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Total Population | Cirrhotics | Poor Responders | Late Responders | Early Responders | Others
Number analyzed (Participants) | 164 | 20 | 24 | 24 | 78 | 18
percentage of participants | 6 [3 to 11] | 5 [0 to 25] | 17 [5 to 37] | 4 [0 to 21] | 0 [0 to 5] | 22 [6 to 48]

9. Secondary Outcome: Percentage of Participants With Treatment Discontinued Based Upon Elevated (Week 12) or Detectable (Week 24) HCV RNA
Description: Treatment was to be discontinued for participants who met prespecified criteria, termed the futility rule, after 12 or 24 weeks of treatment. Participants were discontinued from treatment for one of the following reasons: HCV RNA viral load ≥100 IU/mL (Week 12) or a detectable HCV RNA viral load (Week 24). HCV RNA viral load was measured using the Roche COBAS TaqMan 2.0 HCV Test, with a lower LOD of 10 to 15 IU/mL. The percentage of participants with treatment discontinued for each reason was calculated as [number of participants meeting one of the above criteria divided by the number of participants analyzed] multiplied by 100.
Time Frame: At 12 and 24 weeks
Population: All-Treated Population. Arms were not mutually exclusive.
Measure: Number; unit: percentage of participants
Arm/Group | Total Population | Cirrhotics | Poor Responders | Late Responders | Early Responders | Others
Number analyzed (Participants) | 165 | 20 | 24 | 24 | 78 | 19
percentage of participants
  Week 12 | 4 | 10 | 13 | 0 | 0 | 11
  Week 24 | 3 | 5 | 8 | 0 | 0 | 11

10. Secondary Outcome: Duration of Treatment With PEG-IFN, RBV, and Boceprevir
Description: The duration of treatment with each study drug was determined as the time from treatment start until the last dose of PEG-IFN, RBV, or boceprevir. Median duration of treatment was determined using the actual duration of treatment among individual participants and expressed in weeks.
Time Frame: Up to 48 weeks (from Baseline until EOT)
Population: Safety Population: All participants who received at least one dose of study medication and had at least one post-baseline safety assessment; n = number of participants who received the respective study medication. Arms were not mutually exclusive.
Measure: Median (Full Range); unit: weeks
Arm/Group | Total Population | Cirrhotics | Poor Responders | Late Responders | Early Responders | Others
Number analyzed (Participants) | 165 | 20 | 24 | 24 | 78 | 19
weeks
  PEG-IFN (n=165,20,24,24,78,19) | 28.0 [1 to 49] | 48.0 [14 to 48] | 48.0 [13 to 49] | 48.0 [32 to 48] | 28.0 [24 to 32] | 26.0 [1 to 48]
  RBV (n=165,20,24,24,78,19) | 28.0 [1 to 49] | 48.0 [13 to 48] | 48.0 [14 to 49] | 48.0 [30 to 49] | 28.0 [10 to 33] | 27.0 [1 to 48]
  Boceprevir (n=164,20,24,24,78,18) | 24.0 [1 to 45] | 44.0 [8 to 44] | 44.0 [10 to 45] | 32.0 [2 to 33] | 24.0 [6 to 25] | 10.0 [1 to 44]

11. Secondary Outcome: Percentage of Participants With a Dose Modification of PEG-IFN, RBV, or Boceprevir By Reason
Description: Dose modifications for each study drug included any dose reduction, treatment interruption, or premature withdrawal. Adverse event (AE)-related reasons were documented, as well as reasons related to insufficient efficacy ('Poor efficacy') or other safety-related reasons ('Safety/other'). The percentage of participants with a dose modification documented for each reason was calculated as [number of participants with dose modification divided by the number of participants analyzed] multiplied by 100.
Time Frame: Up to 48 weeks (from Baseline until EOT)
Population: Safety Population; n = number of participants who received the respective study medication. Arms were not mutually exclusive.
Measure: Number; unit: percentage of participants
Arm/Group | Total Population | Cirrhotics | Poor Responders | Late Responders | Early Responders | Others
Number analyzed (Participants) | 165 | 20 | 24 | 24 | 78 | 19
percentage of participants
  PEG-IFN, Any reason (n=165,20,24,24,78,19) | 52 | 60 | 54 | 46 | 42 | 84
  PEG-IFN, Anemia (n=165,20,24,24,78,19) | 1 | 0 | 0 | 0 | 1 | 5
  PEG-IFN, Asthenia (n=165,20,24,24,78,19) | 1 | 0 | 4 | 4 | 0 | 0
  PEG-IFN, Nausea/vomiting (n=165,20,24,24,78,19) | 0.6 | 0 | 0 | 0 | 1 | 0
  PEG-IFN, Neutropenia (n=165,20,24,24,78,19) | 36 | 30 | 38 | 33 | 36 | 47
  PEG-IFN, Rash (n=165,20,24,24,78,19) | 0.6 | 5 | 0 | 0 | 0 | 0
  PEG-IFN, Thrombocytopenia (n=165,20,24,24,78,19) | 5 | 35 | 4 | 0 | 1 | 0
  PEG-IFN, Safety/other (n=165,20,24,24,78,19) | 4 | 10 | 4 | 13 | 0 | 0
  PEG-IFN, Poor efficacy (n=165,20,24,24,78,19) | 8 | 15 | 21 | 4 | 0 | 21
  PEG-IFN, Not specified (n=165,20,24,24,78,19) | 12 | 0 | 8 | 13 | 8 | 42
  RBV, Any reason (n=165,20,24,24,78,19) | 64 | 65 | 67 | 46 | 62 | 89
  RBV, Anemia (n=165,20,24,24,78,19) | 46 | 50 | 46 | 38 | 53 | 26
  RBV, Asthenia (n=165,20,24,24,78,19) | 0.6 | 0 | 0 | 0 | 1 | 0
  RBV, Nausea/vomiting (n=165,20,24,24,78,19) | 1 | 0 | 0 | 0 | 0 | 11
  RBV, Neutropenia (n=165,20,24,24,78,19) | 3 | 0 | 0 | 4 | 0 | 21
  RBV, Rash (n=165,20,24,24,78,19) | 1 | 5 | 0 | 0 | 0 | 5
  RBV, Safety/other (n=165,20,24,24,78,19) | 8 | 15 | 8 | 13 | 3 | 16
  RBV, Poor efficacy (n=165,20,24,24,78,19) | 8 | 15 | 21 | 4 | 0 | 21
  RBV, Not specified (n=165,20,24,24,78,19) | 11 | 0 | 8 | 8 | 8 | 42
  Boceprevir, Any reason (n=164,20,24,24,78,18) | 28 | 45 | 29 | 21 | 12 | 89
  Boceprevir, Anemia (n=164,20,24,24,78,18) | 2 | 10 | 0 | 4 | 0 | 0
  Boceprevir, Asthenia (n=164,20,24,24,78,18) | 0.6 | 0 | 0 | 0 | 1 | 0
  Boceprevir, Nausea/vomiting (n=164,20,24,24,78,18) | 1 | 0 | 0 | 0 | 0 | 11
  Boceprevir, Neutropenia (n=164,20,24,24,78,18) | 4 | 0 | 0 | 4 | 0 | 28
  Boceprevir, Rash (n=164,20,24,24,78,18) | 1 | 5 | 0 | 0 | 0 | 6
  Boceprevir, Safety/other (n=164,20,24,24,78,18) | 4 | 10 | 0 | 4 | 0 | 17
  Boceprevir, Poor efficacy (n=164,20,24,24,78,18) | 7 | 15 | 21 | 0 | 0 | 17
  Boceprevir, Not specified (n=164,20,24,24,78,18) | 12 | 10 | 8 | 8 | 10 | 28

12. Secondary Outcome: Percentage of Participants Receiving Target Administrations of PEG-IFN, RBV, and Boceprevir
Description: The frequency of missed treatments was examined using the number of administrations received as a percentage of target administrations for each study drug. The maximum number of possible administrations was considered in terms of once-weekly injections with PEG-IFN and in terms of treatment days with RBV and boceprevir. The percentage of target administrations each participant received was separated into ranges of <60%, 60 to <80%, 80 to <95%, and ≥95% for each study drug. The percentage of participants who received each range of target administrations was calculated as [number of participants in each range divided by the number of participants analyzed] multiplied by 100.
Time Frame: Up to 48 weeks (from Baseline until EOT)
Population: Safety Population; only participants providing evaluable data were included in the analysis. Arms were not mutually exclusive.
Measure: Number; unit: percentage of participants
Arm/Group | Total Population | Cirrhotics | Poor Responders | Late Responders | Early Responders
Number analyzed (Participants) | 146 | 20 | 24 | 24 | 78
percentage of participants
  PEG-IFN, <60% | 8 | 25 | 25 | 0 | 0
  PEG-IFN, 60 to <80% | 0.7 | 0 | 0 | 4 | 0
  PEG-IFN, 80 to <95% | 5 | 5 | 0 | 17 | 4
  PEG-IFN, 95% or more | 86 | 70 | 75 | 79 | 96
  RBV, <60% | 9 | 25 | 25 | 4 | 1
  RBV, 60 to <80% | 0.7 | 0 | 0 | 4 | 0
  RBV, 80 to <95% | 5 | 10 | 0 | 8 | 4
  RBV, 95% or more | 86 | 65 | 75 | 83 | 95
  Boceprevir, <60% | 10 | 30 | 25 | 8 | 1
  Boceprevir, 60 to <80% | 0.7 | 5 | 0 | 0 | 0
  Boceprevir, 80 to <95% | 3 | 5 | 0 | 4 | 3
  Boceprevir, 95% or more | 86 | 60 | 75 | 88 | 96

13. Secondary Outcome: Number of Participants With a Safety-Related Dose Modification
Description: Dose modifications for each study drug included any dose reduction, treatment interruption, or premature withdrawal. The percentage of participants with a safety-related dose modification (eg, modification due to adverse event or laboratory abnormality) of any study drug was calculated as [number of participants with dose modification divided by the number of participants analyzed] multiplied by 100.
Time Frame: Up to 48 weeks (from Baseline until EOT)
Population: Safety Population.
Measure: Number; unit: participants
Arm/Group | Total Population
Number analyzed (Participants) | 165
participants | 113

14. Secondary Outcome: Time to Safety-Related Dose Modification
Description: Dose modifications for each study drug included any dose reduction, treatment interruption, or premature withdrawal. Median time to safety-related dose modification (eg, modification due to adverse event or laboratory abnormality) of any study drug was estimated using Kaplan-Meier and expressed in weeks.
Time Frame: Up to 48 weeks (from Baseline until EOT)
Population: Safety Population.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Total Population
Number analyzed (Participants) | 165
weeks | 12.1 [10.3 to 16.0]

15. Secondary Outcome: Percentage of Participants Using Concomitant Hematopoietic Stimulants During Treatment and Follow-Up
Description: Use of concomitant hematopoietic stimulants (such as epoetin) during the 48-week treatment period and/or within 24 weeks of follow-up was documented. The percentage of participants using concomitant hematopoietic stimulants was calculated as [number of participants reporting concomitant use divided by the number of participants analyzed] multiplied by 100.
Time Frame: Up to 72 weeks (from Baseline until 24 weeks after EOT)
Population: Safety Population.
Measure: Number; unit: percentage of participants
Arm/Group | Total Population
Number analyzed (Participants) | 165
percentage of participants | 6

16. Secondary Outcome: Percentage of Participants With a Concomitant Disease Prior to or During the Study
Description: The prevalence of concomitant disease at any time from Screening through the end of follow-up was documented. The percentage of participants with a concomitant disease was calculated as [number of participants reporting or diagnosed with concomitant disease divided by the number of participants analyzed] multiplied by 100. Diseases documented for ≥5% of participants included hypertension, diabetes mellitus, hypothyroidism, and vitamin D deficiency as reported here.
Time Frame: Up to 76 weeks (from Screening until 24 weeks after EOT)
Population: Safety Population.
Measure: Number; unit: percentage of participants
Arm/Group | Total Population
Number analyzed (Participants) | 165
percentage of participants
  Any disease | 53
  Hypertension | 18
  Diabetes mellitus | 8
  Hypothyroidism | 6
  Vitamin D deficiency | 5

17. Secondary Outcome: Percentage of Participants Using Concomitant Medications During Treatment and Follow-Up
Description: Use of concomitant prescription or nonprescription medications during the 48-week treatment period and/or within 24 weeks of follow-up was documented. The percentage of participants using concomitant medications was calculated as [number of participants reporting concomitant use divided by the number of participants analyzed] multiplied by 100. Medication classes reported by >10% of participants included analgesics, nonsteroidal anti-inflammatory drugs (NSAIDs), antihistamines, corticosteroids, proton pump inhibitors, vitamins and minerals, and beta-adrenoceptor blocking agents as reported here.
Time Frame: Up to 72 weeks (from Baseline until 24 weeks after EOT)
Population: Safety Population.
Measure: Number; unit: percentage of participants
Arm/Group | Total Population
Number analyzed (Participants) | 165
percentage of participants
  Any medication | 79
  Analgesics | 29
  NSAIDs | 22
  Antihistamines | 19
  Corticosteroids | 19
  Proton pump inhibitors | 17
  Vitamins and minerals | 12
  Beta-adrenoceptor blocking agents | 11

ADVERSE EVENTS:
Time Frame: Up to 72 weeks (from Baseline until 24 weeks after EOT)
Description: Safety Population. Participants were grouped by cirrhotic and noncirrhotic status for the safety analysis, regardless of response-guided treatment rules. Therefore, 21 participants were included in the Cirrhotics (Safety) arm to include one additional participant with cirrhosis who did not fulfill response-guided treatment criteria.
Groups:
- Cirrhotics (Safety): Treatment-naive participants with CHC received treatment with PEG-IFN 180 mcg SC once weekly, weight-based RBV 1000 to 1200 mg PO daily in 2 divided doses, and boceprevir 800 mg PO every 7 to 9 hours. Participants received dual therapy with PEG-IFN and RBV from Week 0 to 4, and triple therapy was initiated at Week 4. Those with undetectable HCV RNA at Weeks 8 and 24 stopped treatment at Week 28. Those with detectable HCV RNA at Week 8 but undetectable HCV RNA at Week 24 continued triple therapy until Week 36 and received dual therapy from Week 36 to 48. Those with a <1-log decrease in HCV RNA at Week 4 continued triple therapy until Week 48, with optional dual therapy from Week 32 to 48 if triple therapy was not tolerated. Participants with compensated cirrhosis, regardless of response, received triple therapy until Week 48. Participants with liver cirrhosis were grouped separately in the safety analysis.
- Noncirrhotics (Safety): Treatment-naive participants with CHC received treatment with PEG-IFN 180 mcg SC once weekly, weight-based RBV 1000 to 1200 mg PO daily in 2 divided doses, and boceprevir 800 mg PO every 7 to 9 hours. Participants received dual therapy with PEG-IFN and RBV from Week 0 to 4, and triple therapy was initiated at Week 4. Those with undetectable HCV RNA at Weeks 8 and 24 stopped treatment at Week 28. Those with detectable HCV RNA at Week 8 but undetectable HCV RNA at Week 24 continued triple therapy until Week 36 and received dual therapy from Week 36 to 48. Those with a <1-log decrease in HCV RNA at Week 4 continued triple therapy until Week 48, with optional dual therapy from Week 32 to 48 if triple therapy was not tolerated. Participants with compensated cirrhosis, regardless of response, received triple therapy until Week 48. Participants without liver cirrhosis, including those with transition to cirrhosis, were grouped separately in the safety analysis.
Arm/Group | Cirrhotics (Safety) | Noncirrhotics (Safety)
Serious Adverse Events (participants affected / at risk) | 7/21 | 8/144
Other Adverse Events (participants affected / at risk) | 21/21 | 135/144
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cirrhotics (Safety) (N=21) | Noncirrhotics (Safety) (N=144)
Anaemia (Blood and lymphatic system disorders) | 2 | 2
Granulocytopenia (Blood and lymphatic system disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Fatigue (General disorders) | 0 | 1
Hepatic failure (Hepatobiliary disorders) | 2 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1
Hepatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 1
Epididymitis (Infections and infestations) | 0 | 1
Depression (Psychiatric disorders) | 0 | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cirrhotics (Safety) (N=21) | Noncirrhotics (Safety) (N=144)
Asthenia (General disorders) | 7 | 40
Influenza like illness (General disorders) | 6 | 34
Fatigue (General disorders) | 4 | 31
Pyrexia (General disorders) | 0 | 26
Neutropenia (Blood and lymphatic system disorders) | 5 | 47
Anaemia (Blood and lymphatic system disorders) | 7 | 57
Thrombocytopenia (Blood and lymphatic system disorders) | 6 | 13
Dysgeusia (Nervous system disorders) | 6 | 45
Headache (Nervous system disorders) | 2 | 32
Dizziness (Nervous system disorders) | 1 | 13
Somnolence (Nervous system disorders) | 2 | 4
Pruritus (Skin and subcutaneous tissue disorders) | 4 | 30
Rash (Skin and subcutaneous tissue disorders) | 3 | 19
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 19
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 8
Erythema (Skin and subcutaneous tissue disorders) | 2 | 5
Nausea (Gastrointestinal disorders) | 3 | 23
Diarrhoea (Gastrointestinal disorders) | 4 | 15
Dyspepsia (Gastrointestinal disorders) | 3 | 11
Vomiting (Gastrointestinal disorders) | 1 | 8
Abdominal pain (Gastrointestinal disorders) | 0 | 9
Gastritis (Gastrointestinal disorders) | 2 | 2
Stomatitis (Gastrointestinal disorders) | 2 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 13
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 13
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 31
Insomnia (Psychiatric disorders) | 3 | 17
Decreased appetite (Metabolism and nutrition disorders) | 1 | 13
Weight decreased (Investigations) | 2 | 8
Hypertension (Vascular disorders) | 2 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.